CLINICAL TRIAL: NCT03679572
Title: Zero-ischemia Robot-assisted Partial Nephrectomy Using Near-infrared Fluorescence: A Prospective, Monocentric, Randomized, Comparative and Open-label Study
Brief Title: Zero-ischemia Robot-assisted Partial Nephrectomy Using Near-infrared Fluorescence
Acronym: EMERALD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC17.142
Record Dates: First submitted 2018-03-26; First posted 2018-09-20 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Renal Cancer
Keywords: partial nephrectomy; robot-assisted; surgery; near-infrared fluorescence; ischemia
MeSH Terms: conditions — Kidney Neoplasms; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot assisted partial nephrectomy super-selective clamping (Experimental): The Da Vinci robot (device) allows to use near-infrared fluorescence in order to clamp precisely the branches of the vascularization for the partial nephrectomy. The healthy parenchyma ischemia is avoided.
  Interventions: Procedure: Robot assisted partial nephrectomy super-selective clamping
- Robot assisted partial nephrectomy with renal artery clamping (Active Comparator): The partial nephrectomy with robotic assistance is performed using a renal artery. It's the conventional method.
  Interventions: Procedure: Robot assisted partial nephrectomy with renal artery clamping

INTERVENTIONS:
Procedure: Robot assisted partial nephrectomy super-selective clamping — The device used to performe the surgery is a Da Vinci robot. After injection of infracyanine, the super-selective clamping is possible. The surgery is performed using a specific clamping of the tumor arteries. Super-selective ischemia is checked using near infrared fluorescence.
  Other Names: Robot assisted zero-ischemia partial nephrectomy with the Da Vinci robot (device)
  Arms: Robot assisted partial nephrectomy super-selective clamping
Procedure: Robot assisted partial nephrectomy with renal artery clamping — Partial nephrectomy is performed with the conventional method in wich a renal artery clamping is done.
  Other Names: Robot assisted partial nephrectomy with conventional method
  Arms: Robot assisted partial nephrectomy with renal artery clamping

SUMMARY:
Patients with renal cancer are commonly treated by robot-assisted partial nephrectomy. Renal artery clamping is commonly required inducing kidney ischemia during surgery. It impacts parenchymal and renal function. This study aims to compare a new surgical procedure in order to reduce ischemia effect and preserve renal function after partial nephrectomy for renal tumour.

ELIGIBILITY:
Inclusion Criteria:

* candidate for a robot-assisted partial nephrectomy for renal tumour
* patient affiliated to social security
* signature of the informed consent

Exclusion Criteria:

* proven or suspected allergy to the indocyanine green
* coagulation disorder contraindicating robot assistance in the partial nephrectomy
* medical pathology contraindicating pneumo-peritoneum
* multiple tumors
* horseshoe kidney
* exclusion period of another interventionnal study
* protected person referred to in Articles L1121-5 to L1121-8 of the Code of Public Health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Benefit on postoperative renal function of fluorescence-enhanced super-selective clamping during robot assisted partial nephrectomy compared with robot-assisted partial nephrectomy with renal artery clamping | 6 months
  The glomerular filtration rate (GFR) of the kidney operated is assessed at 6 months after surgery. This value is compared to that assessed before the surgery to see the variation. This variation is compare between the two groups.

SECONDARY OUTCOMES:
Number of group conversion in the zero ischemia method. | 6 months
  The feasibility of the new technique is assessed by counting the number of group conversion towards conventional technique.
Surgical duration in the two groups | 6 months
  Duration between the first incision and the skin closure
Complications | 1 month
  number of complications per and post-surgery up to 1 month
Per-surgery blood loss | 1 month
  per-surgery blood loss in millimeter
Hemoglobine rate variation | 1 month
  For patients having no received blood transfusion, the hemoglobine rate variation is assessed in percentage at one month in post-surgery.
Positive surgical margins | 1 month
  Number of positive surgical margins
Variation between global GFR in the two groups | 6 months
  The variation of the global GFR is assessed after surgery, when patient is discharged. This value is compared to the that collected before the surgery.
Renal parenchyma preserved | 6 months
  The percentage of renal parenchyma preserved is evaluated by CT renal volumetry at 6 months after the surgery. The value is compared to that collected before the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Alexandre Long, MD, PhD, Principal Investigator — department of urology and renal transplantation
Locations (1):
- University Hospital Grenoble-Alps (CHU-GA), La Tronche, France

REFERENCES:
- [Derived] Long JA, Fiard G, Giai J, Teyssier Y, Fontanell A, Overs C, Poncet D, Descotes JL, Rambeaud JJ, Moreau-Gaudry A, Ittobane T, Bouzit A, Bosson JL, Lanchon C. Superselective Ischemia in Robotic Partial Nephrectomy Does Not Provide Better Long-term Renal Function than Renal Artery Clamping in a Randomized Controlled Trial (EMERALD): Should We Take the Risk? Eur Urol Focus. 2022 May;8(3):769-776. doi: 10.1016/j.euf.2021.04.009. Epub 2021 Apr 27. PMID 33931361